CLINICAL TRIAL: NCT03091933
Title: An Exploratory, Open-label, Multicenter Study to Evaluate the Safety and Efficacy of Anti-minor Histocompatibility Complex (MiHA) Donor T-lymphocytes Expanded ex Vivo, in Patients With a Hematologic Malignancy, With Molecular or Clinical Relapse After Hematopoietic Stem Cell Transplantation From a Matched Donor
Brief Title: Antiminor Histocompatibility Complex (MiHA) T Cells for Patients With Relapsed Hematologic Malignancies Following Matched HSCT (Guided Lymphocyte Immunopeptide Derived Expansion)
Acronym: GLIDE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-MIHA-001
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Hematologic Cancer; Relapse Leukemia; Relapsed Adult ALL; Relapsed Adult AML; Relapsed CLL; Relapsed Non Hodgkin Lymphoma; Relapsed Hodgkin's Lymphoma; Relapsed Myelodysplastic Syndromes; Relapsed Multiple Myeloma
Keywords: allogeneic hematopoietic stem cell transplantation; relapsed hematopoietic malignancy; HLA matched donor; minor histocompatibilty antigen (MiHA)
MeSH Terms: conditions — Hematologic Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Hodgkin Disease; Myelodysplastic Syndromes; Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: exploratory, open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GLIDE (Experimental): GLIDE single infusion at a target dose of 4x107 viable T-cells/m2
  Interventions: Biological: GLIDE

INTERVENTIONS:
Biological: GLIDE — Gudide Lymphocyte by Immunopeptide Derived Expansion (GLIDE) is an anti- Minor histocompatibility (MiHA) cell line

SUMMARY:
This study will evaluate the safety of infusing an anti-MiHA T cell line in patients suffering from an hematologic malignancy that has relapsed following hematopoietic stem cell transplantation from a matched donor.

DETAILED DESCRIPTION:
The GLIDE-201/44 trial primarily aims to test the safety of anti-MiHA T cell line in patients suffering from an hematologic malignancy that has relapsed following hematopoietic stem cell transplantation from a matched donor. The anti-MiHA T cell lines are derived from the matched donor for the patient, the original donor for a given patient. Both the patient and the matched donor will undergo screening to determine the expression of targetable MiHAs. Upon identification of the target MiHAs, donor cells will be collected through apheresis and primed against the selected MiHA. In this setting, the GLIDE 201/44 product will be cryopreserved, thawed and administered as a single infusion at a target dose of 4x10E+07 viable T cells/m2 (range of dose is 0.4 4x10E+07 viable T cells/m2). A second infusion can be offered to the patients after an observation period of 42 days upon clinical evaluation by the treating physician. In the absence of secondary adverse events following the initial infusion, a second infusion of the GLIDE 201/44 product could be administered at a dose level up to 3-5 fold the original dose.

ELIGIBILITY:
Inclusion Criteria:

* Prior allogeneic HLA-matched stem cell transplantation
* Any of the following hematologic malignancies:
* Acute myeloid leukemia (AML)
* Acute lymphoblastic leukemia (ALL)
* Biphenotypic leukemia
* Chronic lymphoblastic leukemia (CLL)
* Hodgkin Lymphoma
* Non-Hodgkin Lymphoma (NHL)
* Multiple Myeloma (MM)
* Myelodysplastic syndrome (MDS)
* Presence of HLA2:01 and / or HLA44:02 and / or HLA-B*44:03, HLA-A*01:01; HLA-A*03:01; HLA-A*11:01;HLA A*24:02; HLA-A*29:02; HLA-A*32:01; HLA-B*07:02; HLA-B*08:01; HLA B*13:02; HLA-B*14:02; HLA-B*15:01; HLA-B*18:01; HLA-B*27:05; HLA B*35:01; HLA-B*40:01; or HLA-B*57:01
* At least 6 months after allogeneic hematopoietic stem cell transplantation
* Presence of detectable malignant disease post-transplantation in the form of molecular, cytogenetic or hematologic relapse of the malignant disorder.
* Eligible to receive cytoreductive chemotherapy
* Original stem cell donor available for leukocyte donation.
* ECOG performance status ≤2.
* Ability to provide written consent.
* Accessible for treatment and follow up.
* Presence of a targetable MiHA based on exome sequencing of the patient and donor

Exclusion Criteria:

* Active acute GVHD > grade I
* Prior grade III-IV acute GVHD within the last year
* Uncontrolled chronic GVHD
* Prior administration of donor lymphocyte infusion (DLI)
* Use of T-cell depleting antibodies in the previous 30 days
* Treatment with immune suppressors (oral or parenteral steroids corresponding to a dose of prednisone greater than 7.5 mg/day, calcineurine inhibitors, rapamycin, mycophenolate mofetil, etc) during the last 30 days.
* Uncontrolled active infection
* Uncontrolled central nervous system involvement by leukemia cells (blasts).
* AST or ALT > 2.5 x ULN (CTCAE grade 2)
* Bilirubin > 1.5 x ULN (CTCAE grade 2)
* Creatinine clearance < 50 mL/min
* Positive test for human immunodeficiency virus (HIV)
* Positive pregnancy test (women of childbearing age only)
* Lactating women: the safety of this therapy on breast milk is not known.
* Estimated probability of surviving less than 3 months
* Known allergy to any of the components of GLIDE (e.g., dimethyl sulfoxide)
* Intercurrent illness or medical condition precluding safe administration of the planned protocol treatment or required follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-02-06 (Actual); Primary Completion 2018-03-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Non-hematologic toxicity related to GLIDE post injection | 6 months
  No death or other toxic events directly related to GLIDE injection

SECONDARY OUTCOMES:
Response of hematologic malignancy (acute leukemia (ALL, AML, biphenotypic), CLL, HL, NHL, MM or MDS) post-injection | up to 12 months
  Disease progression following GLIDE injection
Incidence and severity of acute and chronic graft versus host disease (GvHD) | up to 12 months
  Progression (if any) or induction of GvHD
Persistence of GLIDE in the host and homing to peripheral blood, bone marrow and other tissues | up to 12 months
  Monitoring of GLIDE product persistence in host
Non-Relapse mortality (NRM) | up to 12 months
  Time to deaths without relapse/recurrence
Relapse-incidence (RI) | up to 12 months
  Time to relapse
Overall survival (OS) | up to 12 months
  Time to death, irrespective of the cause
Progression-free survival (PFS) | up to 12 months
  It is time to any of the following: OS, RI, NRM, Time to relapse, Relapse free survival

CONTACTS AND LOCATIONS:
Overall Officials: Denis-Claude Roy, MD PhD, Principal Investigator — CIUSSS d l'Est-de-l'Île-de-Montréal; Jean-Sébastien Delisle, MD PhD, Principal Investigator — CIUSSS d l'Est-de-l'Île-de-Montréal; Silvy Lachance, MD, Principal Investigator — CIUSSS d l'Est-de-l'Île-de-Montréal
Locations (1):
- CIUSSS d l'Est-de-l'Île-de-Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data for all primary and secondary outcome measures will be made available within 6 months of study end